CLINICAL TRIAL: NCT02139436
Title: Hybrid-FES Exercise to Prevent Cardiovascular Declines in Acute SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, J. Andrew Taylor, Director, Cardiovascular Research Laboratory, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R01HL117037 (NIH); 1R01HL117037 (NIH)
Record Dates: First submitted 2014-05-12; First posted 2014-05-15 (Estimated); Results first posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-02

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Flowering time control protein FCA, Arabidopsis

STUDY DESIGN:
Intervention Model Description: Three intervention groups (Control, AO-Row, and FES-RT) run in parallel
Oversight: Data Monitoring Committee: No

ARMS (3):
- FES-row-training (Experimental): Subjects will perform 6 months of FES-row-training.
  Interventions: Other: FES-row-training
- Wait-list time control (Other): Subjects perform 6 months of their standard of care
  Interventions: Other: Time Control
- Arms-only-row-training (Active Comparator): Subjects will perform 6 months of arms-only row training
  Interventions: Other: Arms-only-row training

INTERVENTIONS:
Other: FES-row-training
  Arms: FES-row-training
Other: Arms-only-row training
  Arms: Arms-only-row-training
Other: Time Control
  Arms: Wait-list time control

SUMMARY:
Each year, 11,000 people suffer a spinal cord injury (SCI) in the U.S. Within the first year, there are profound declines in physiologic function, forming the underlying substrate for future cardiovascular disease . In fact, acquired cardiovascular disease is an increasingly recognized consequence of SCI and is the leading cause of death in SCI. Though incompletely understood, the almost 10-fold prevalence of cardiovascular disease results in part from profound physiologic 'detraining' resulting from motor impairment and immobility. Currently, effective interventions preventing acute declines that lead to cardiovascular compromise and increased risk in SCI are lacking - exercise therapy for those with SCI is challenging and when employed, is typically limited to the upper body. Recently, the investigators refined a unique form of exercise for those with SCI that specifically mirrors exercise performed by those without SCI. Functional Electrical Stimulation (FES) Row Training (RT) couples volitional arm and electrically controlled leg exercise, resulting in a hemodynamic profile that produces the beneficial cardiac loading conditions of large muscle mass exercise. As such, FES-RT may be a safe and effective way to attenuate cardiovascular declines following SCI. The investigators aims are to test the overall hypotheses that FES-RT will: 1) mitigate against increased visceral adiposity and reduced insulin sensitivity, 2) prevent worsening lipid profile and compromised baroreflex function, and 3) counter ventricular wall thickening and declining ventricular function occurring with acute SCI, and that these effects will be greater than that observed with an arms-only exercise group. Changes with FES-RT will be compared to a time (wait-list) control and to arms-only-RT. Individuals with an SCI within the last 3-6 months will be randomized to FES-RT, to a time control, or arms-only-RT. Measures will be made at baseline and 6 months. The investigators work will provide results that clearly delineate potential health benefits of FES-RT, and if FES-RT is effective in a majority of those with SCI, its application, implementation, and integration could be easily replicated.

DETAILED DESCRIPTION:
We will enroll approximately 60 individuals within three to six months post SCI to obtain data on 50 individuals. One-half of the subjects (N=25) will be randomized to immediately enroll in 6 months of FES-RT. One third (N=18) will be randomized to a wait-list to provide time control data from baseline to 6 months. A wait-list control group is routine in exercise studies because most volunteers are interested in participating in an exercise program. Hence, time controls are difficult to capture since many of those randomized to receive no exercise either drop from the study entirely, or end up pursuing some form of exercise on their own. Therefore, a vehicle for enrollment of a time control group that is acceptable to most volunteers is a wait-list. Therefore, a six month time control will provide data on expected declines and then subjects will be randomized to six months exercise.

Training Protocols for Each Study Group

1. FES-RT GROUP

   Subjects will begin with short intervals of FES-RT interspersed with rest intervals and/or arms-only rowing intervals depending on fitness level and the response to the FES. A maximum FES-rowing test will be performed at baseline. This will be repeated after three months of training and training intensity will be adjusted to maintain the training stimulus at the same relative intensity. The goal is for each volunteer to achieve an exercise intensity of 75-85% maintained for a continuous 30 minutes performed three times each week. A maximum FES-rowing test will be performed at the end of the six months of FES-RT to determine increases in fitness.
2. ARMS-ONLY-RT GROUP

   Training sessions will be 3 times per week for 26 weeks. To parallel the FES-RT, the initial training sessions will also consist of 6 sets of arms-only rowing for five minutes at 60% of VO2peak with a work-to-rest ratio of 2:1 and progress over the six months to an exercise intensity of 75-85% maintained for 30 minutes performed three times each week. A maximum arms-only rowing test will be performed at baseline. This will be repeated after three months of training and training intensity will be adjusted to maintain the training stimulus at the same relative intensity. A maximum arms-only rowing test will be performed at the end of the six months of training to determine increases in fitness.
3. WAIT-LIST GROUP

The wait list group will not participate in any training for 6 months. A maximum arms-only rowing test will be performed immediately after enrollment, after initial familiarization with arms-only-RT equipment (usually 2-3 sessions) and will be repeated after 3 and 6 months

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injured outpatients aged 18-40
* medically stable
* body mass index 18.5-30.0
* 3-12 months post SCI
* ASIA scale A, B or C at neurological level C5-T12
* able to follow directions
* leg muscles responsive to FES

Exclusion Criteria:

* hypertension
* significant arrhythmias
* coronary artery disease
* diabetes
* renal disease
* cancer
* epilepsy
* current use of cardioactive medications
* current grade 2 or greater pressure ulcers at relevant contact sites
* other neurological disease
* peripheral nerve compressions or rotator cuff tears that limit ability to row
* history of bleeding disorder

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2013-12; Primary Completion 2020-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Andrew Taylor, Ph.D., Principal Investigator — Spaulding Rehabilitation Hospital/Harvard Medical School
Locations (1):
- Spaulding Hospital Cambridge, Cambridge, Massachusetts, United States

REFERENCES:
- [Derived] Yates BA, Brown R, Picard G, Taylor JA. Improved pulmonary function is associated with reduced inflammation after hybrid whole-body exercise training in persons with spinal cord injury. Exp Physiol. 2023 Mar;108(3):353-360. doi: 10.1113/EP090785. Epub 2023 Jan 9. PMID 36622954
- [Derived] Ely MR, Schleifer GD, Singh TK, Baggish AL, Taylor JA. Exercise Training Does Not Attenuate Cardiac Atrophy or Loss of Function in Individuals With Acute Spinal Cord Injury: A Pilot Study. Arch Phys Med Rehabil. 2023 Jun;104(6):909-917. doi: 10.1016/j.apmr.2022.12.001. Epub 2022 Dec 23. PMID 36572202
- [Derived] Solinsky R, Schleifer GD, Draghici AE, Hamner JW, Taylor JA. Methodologic implications for rehabilitation research: Differences in heart rate variability introduced by respiration. PM R. 2022 Dec;14(12):1483-1489. doi: 10.1002/pmrj.12770. Epub 2022 Mar 12. PMID 35077032
- [Derived] Solinsky R, Draghici A, Hamner JW, Goldstein R, Taylor JA. High-intensity, whole-body exercise improves blood pressure control in individuals with spinal cord injury: A prospective randomized controlled trial. PLoS One. 2021 Mar 4;16(3):e0247576. doi: 10.1371/journal.pone.0247576. eCollection 2021. PMID 33661958
- [Derived] Ely MR, Singh TK, Baggish AL, Taylor JA. Reductions in Cardiac Structure and Function 24 Months After Spinal Cord Injury: A Cross-Sectional Study. Arch Phys Med Rehabil. 2021 Aug;102(8):1490-1498. doi: 10.1016/j.apmr.2021.01.070. Epub 2021 Feb 5. PMID 33556347

RESULTS

PARTICIPANT FLOW:
Groups:
- FES-row-training: Subjects will perform 6 months of FES-row-training.
  FES-row-training
- Wait-list Time Control: Subjects perform 6 months of their standard of care
  Time Control
- Arms-only-row-training: Subjects will perform 6 months of arms-only row training
  Arms-only-row training
Period: Overall Study
Arm/Group | FES-row-training | Wait-list Time Control | Arms-only-row-training
Started | 41 | 14 | 13
Completed | 41 | 14 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis is a subset of the total number of participants in the whole study from which complete data was available
Groups:
- Total: Total of all reporting groups
Arm/Group | FES-row-training | Wait-list Time Control | Arms-only-row-training | Total
Number analyzed (Participants) | 41 | 14 | 13 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 41 | 14 | 13 | 68
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (5) | 28 (6) | 28 (6) | 28 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 1 | 10
  Male | 33 | 13 | 12 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 3 | 7
  White | 28 | 11 | 8 | 47
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 6 | 0 | 1 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 14 | 13 | 68

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Exercise Capacity at 6 Months
Description: Volunteers will perform an incremental exercise test of FES- or arms-only rowing to determine maximal oxygen uptake.
Time Frame: Baseline and 6 months
Population: The reported results represent a sub-population of the total number of subjects who completed the study. Some subjects did not complete the 6 month VO2 or their results were removed due to quality control or not meeting the criteria for a good test. Therefore, the presented numbers represent reliable and unbiased data.
Measure: Mean (Standard Error); unit: ml/kg/min
Groups:
- Waitlist Controls: Controls (no structured exercise)
- Arms Only: Arms Only Rowing
- FES-Rowing: Functional Electrical Stimulation Rowing
Arm/Group | Waitlist Controls | Arms Only | FES-Rowing
Number analyzed (Participants) | 11 | 11 | 16
ml/kg/min
  Baseline | 14.6 (3.4) | 18.5 (3.7) | 17.1 (1.2)
  6 Months | 13.9 (2.5) | 18.2 (4.4) | 18.9 (1.5)

2. Primary Outcome: Change From Baseline in Visceral Adiposity at 6 Months
Description: We will use a 5th generation General Electric Healthcare dual x-ray absorptiometry(DXA) scanner for regional fat measurements, the DXA software can be used to define standard regions that will allow comparability of measurements throughout the study.
Time Frame: Baseline, 6 months
Population: These are subgroups of the main study population. Exercise groups were combined.
Measure: Mean (Standard Error); unit: g
Groups:
- Waitlist: Subjects continued with standard of care and did not perform and structured exercise
- FES Rowing: Subjects that performed FES-rowing
- Arms-Only Rowing: Subjects that only performed Arms-only rowing
Arm/Group | Waitlist | FES Rowing | Arms-Only Rowing
Number analyzed (Participants) | 6 | 18 | 7
g
  Baseline | 13649 (1320) | 10503 (1235) | 10945 (2310)
  6-Months | 16057 (1952) | 11247 (1390) | 12197 (2492)

3. Primary Outcome: Change From Baseline in Myocardial Structure at 6 Months.
Description: Echocardiography was performed using a commercially available system(Vivid-1, General Electric Healthcare)to obtain measures of left ventricular wall thickness and left ventricular diastolic function.
Time Frame: Baseline and 6 months
Population: The reported results represent a sub-population of the total number of subjects who completed the study. Some subjects did not complete the 6 month echocardiography or their results were removed due to quality control or not meeting the criteria for a good test. Therefore, the presented numbers represent reliable and unbiased data.
Measure: Mean (Standard Error); unit: g
Arm/Group | Waitlist Controls | Arms Only | FES-Rowing
Number analyzed (Participants) | 7 | 6 | 17
g
  Baseline | 136 (4) | 149 (5) | 143 (2)
  6 Months | 129 (8) | 133 (4) | 138 (4)

4. Primary Outcome: Change From Baseline in Insulin Sensitivity at 6 Months.
Description: Blood will be taken via standard venipuncture to measure the homeostasis model assessment of insulin resistance (HOMA-IR). HOMA-IR is a measure of insulin resistance/sensitivity calculated by multiplying fasting insulin (μU/mL) by fasting glucose (mg/dL) and divided by a constant (405). A higher value indicates higher insulin resistance.
Time Frame: Baseline and 6 months
Population: The reported results represent a sub-population of the total number of subjects who completed the study. Some subjects did not complete the 6 month blood draw. Therefore, the presented numbers represent reliable and unbiased data.
Measure: Mean (Standard Error); unit: HOMA-IR Index
Arm/Group | Waitlist Controls | Arms Only | FES-Rowing
Number analyzed (Participants) | 4 | 2 | 16
HOMA-IR Index
  Baseline | 2.7 (1.7) | 0.9 (0.1) | 1.4 (0.5)
  6 Months | 3.1 (1.5) | 0.6 (0.2) | 1.7 (0.6)

5. Primary Outcome: Change From Baseline in Blood Lipids at 6 Months
Description: Blood will be taken via standard venipuncture to measure: total cholesterol.
Time Frame: Baseline and 6 months
Population: as for outcome 4
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | FES-row-training | Wait-list Time Control | Arms-only-row-training
Number analyzed (Participants) | 16 | 4 | 2
mg/dL
  Baseline | 170 (8) | 157 (9) | 158 (4)
  6 Months | 171 (8) | 141 (10) | 149 (4)

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | FES-row-training | Wait-list Time Control | Arms-only-row-training
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/14 | 1/13
Other Adverse Events (participants affected / at risk) | 8/41 | 0/14 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FES-row-training (N=41) | Wait-list Time Control (N=14) | Arms-only-row-training (N=13)
Autonomic Dysreflexia (Cardiac disorders) | 0 (0) | 1 (2) | 1 (2) — Autonomic dysreflexia (AD) characterized by a sudden abnormal elevation in blood pressure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FES-row-training (N=41) | Wait-list Time Control (N=14) | Arms-only-row-training (N=13)
Low Blood Pressure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Low BP is common in individuals with SCI. Excluded from exercise if BP is low.
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) — Pressure ulcers are common in individuals with SCI
Elevated Blood Pressure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Temporary elevations in blood pressure, not related to autonomic dysreflexia, which subsides with 10 minutes of rest
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) — Inflammation of a joint.
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) — Reports of sickness following exercise/testing

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT02139436/Prot_SAP_000.pdf